CLINICAL TRIAL: NCT06873035
Title: A Phase 2/3, Multicenter, Open-Label Phase Followed by a Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Infigratinib in Children With Hypochondroplasia: ACCEL 2/3
Brief Title: An Interventional Study of Infigratinib in Children With Hypochondroplasia
Acronym: HCH
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: QED Therapeutics, a BridgeBio company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QBGJ398-304
Record Dates: First submitted 2025-02-18; First posted 2025-03-12 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-03

CONDITIONS: Hypochondroplasia
Keywords: skeletal dysplasia; endochondral ossification; hypochondroplasia; HCH; shortened proximal limbs; fibroblast growth factor receptor 3; FGFR3; endochondral bone formation; disproportionate short stature; quality of life; dwarfism; bone diseases; musculoskeletal diseases; osteochondrodysplasia; functional abilities; annualized growth velocity; annualized height velocity; growth; genetic diseases; congenital; AHV; AGV; Pathogenic variants
MeSH Terms: conditions — Hypochondroplasia; Mucopolysaccharidosis IV; Dwarfism; Bone Diseases; Musculoskeletal Diseases; Osteochondrodysplasias; Genetic Diseases, Inborn | interventions — infigratinib

STUDY DESIGN:
Intervention Model Description: This study comprises an open-label Phase 2 portion to evaluate safety and efficacy in participants receiving infigratinib at one of two doses followed by a Phase 3 randomized, double-blind portion of the dose selected from the Phase 2 portion versus placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 2 Cohort 1 (Experimental): infigratinib (0.128 mg/kg/day)
  Interventions: Drug: infigratinib 0.128 mg/kg/day
- Phase 2 Cohort 2 (Experimental): infigratinib (0.25 mg/kg/day)
  Interventions: Drug: infigratinib 0.25 mg/kg/day

INTERVENTIONS:
Drug: infigratinib 0.128 mg/kg/day — Oral infigratinib 0.128 mg/kg/day
  Arms: Phase 2 Cohort 1
Drug: infigratinib 0.25 mg/kg/day — Oral infigratinib 0.25 mg/kg/day
  Arms: Phase 2 Cohort 2

SUMMARY:
ACCEL2/3 is a Phase 2/3 study. The purpose of the Phase 2 portion of the study (ACCEL2/3) is to evaluate the efficacy and safety, of infigratinib in children with hypochondroplasia (HCH) receiving infigratinib, at one of two doses, of who have completed at least 26 weeks of participation in QED-sponsored ACCEL (QBGJ398-004).

DETAILED DESCRIPTION:
ACCEL 2/3 is a Phase 2/3 study that comprises of 2 portions. The Phase 2 portion is an open-label, portion in children with HCH aged 5 to 11 years old followed by a Phase 3 portion which is double-blind, placebo-controlled in children with HCH aged >3 years old to <18 years old.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must have completed at least 26 weeks and still be on the observational study (QBGJ398-004).
* Phase 2 portion: Participants 5-11 years of age (inclusive).
* Phase 3 portion: Participants 3 to <18 years of age at screening with growth potential
* Diagnosis of HCH documented clinically by the presence of disproportionate short stature and confirmed with a molecular test.
* Participants are able to swallow oral medication.
* Participants and parent(s), legal guardian(s), or caregiver(s) are willing and able to comply with study visits and study procedures.
* Participants are ambulatory and able to stand without assistance. Sex and Contraceptive/Barrier Requirements
* Negative pregnancy test in girls ≥10 years of age or girls of any age who have experienced menarche.
* If sexually active, participants whether male or female, must be willing to use a highly effective method of contraception, as relevant, while taking study drug and for 1 month after the last dose of study drug.
* Signed informed consent.

Key Exclusion Criteria:

* Participants who have ACH or a short stature condition other than HCH.
* Significant concurrent disease or condition that, in the view of the investigator and/or sponsor, would confound assessment of efficacy or safety of infigratinib.
* Current evidence of clinically significant corneal or retinal disorder/keratopathy confirmed by ophthalmic examination.
* Concurrent circumstance, disease, or condition that, in the view of the investigator and/or sponsor, would interfere with study participation or safety evaluations.
* History and/or current evidence of extensive ectopic tissue calcification.
* History of malignancy.
* Having received or planning to receive treatment with any other investigational or approved product for the treatment of ACH, HCH, or short stature.
* Regular long-term treatment (≥3 weeks) with supraphysiologic doses of glucocorticoid.
* Previous limb-lengthening surgery at any time or planned/expected to have limb-lengthening or guided growth surgery while participating in the study.
* Participants receiving medications which could increase serum phosphorus and/or calcium concentrations
* Clinically significant abnormality in any laboratory test result at screening.
* Pregnant or breastfeeding at the screening visit or planning to become pregnant (self or partner) at any time during the study.
* Allergy to any components of the study drug.
* Concurrent circumstance, disease, or condition that would interfere with study participation.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline (BL) in Annualized Height Velocity (AHV; cm/year) | 26 weeks
Incidence, severity, and seriousness of adverse events (AEs) that require dose reduction or discontinuation | at least 26 weeks

SECONDARY OUTCOMES:
Change from BL in height Z-score (in relation to both HCH and average height tables) | 52 weeks
Change from BL in upper to lower body segment ratio (cm) | 52 weeks
Changes in cognitive function (as assessed by age appropriate computerized tests) | 52 weeks
Pharmacokinetic profile of infigratinib by assessment of maximum concentration (Cmax) | 52 weeks
Pharmacokinetic profile of infigratinib by assessment of time-to-maximum concentration (Tmax) | 52 weeks
Change from BL in collagen X marker (CXM) levels | 52 weeks

OTHER OUTCOMES:
Change from BL in comorbidities associated with HCH | 52 weeks
Change from BL in Health-related Quality of Life (HRQoL) (as assessed by Pediatric Quality of Life Inventory [PedsQL tool]) | 52 weeks
Evaluate treatment benefit as assessed by qualitative interviews | 52 weeks

CONTACTS AND LOCATIONS:
Locations (22):
- United States (7):
  - UCSF Benioff Children's Hospital, Oakland, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Children's National Hospital, Washington D.C., District of Columbia
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - University of Missouri, Columbia, Missouri
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Wisconsin Madison - Waisman Center Bone Dysplasia Clinic, Madison, Wisconsin
- Murdoch Children's Research Institute, Parkville, Victoria, Australia
- Canada (3):
  - London Health Services Center - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario Research Institute, Ottawa, Ontario
  - Université de Montréal - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
- France (3):
  - Hôpital Femme Mère Enfant, Bron, France
  - Hôpital Universitaire Necker-Enfants Malades, Paris, France
  - Centre Hospitalier Universitaire (CHU) de Toulouse - Hôpital des Enfants, Toulouse, France
- Norway (2):
  - Haukeland University Hospital, Bergen, Norway
  - Paediatric Clinical Research Unit at Osla University Hospital, Oslo, Norway
- Hospital Pediátrico de Coimbra, Coimbra, Portugal, Portugal
- KK Women's and Children's Hospital, Singapore, Singapore, Singapore
- Hospital Vithas San Jose, Vitoria-Gasteiz, Spain, Spain
- Astrid Lindgren Children's Hospital, Solna, Sweden, Sweden
- United Kingdom (2):
  - Manchester University, Manchester, United Kingdom
  - Sheffield Children's Hospital, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No